CLINICAL TRIAL: NCT02558790
Title: L-Threonic Acid Magnesium Salt (L-TAMS) in ADHD: An Open-label Pilot Study of Cognitive and Functional Effects
Brief Title: L-Threonic Acid Magnesium Salt (L-TAMS) in ADHD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Neurocentria, Inc. (Industry)
Responsible Party: Principal Investigator, Craig B. Surman, MD, Scientific Coordinator of the Adult ADHD Program, Clinical and Research Program in Pediatric Psychopharmacology and Adult ADHD, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014-P-000528
Record Dates: First submitted 2015-09-23; First posted 2015-09-24 (Estimated); Results first posted 2018-05-14 (Actual); Last update posted 2018-05-14 (Actual); Status verified 2018-04

CONDITIONS: Attention Deficit/Hyperactivity Disorder; ADHD
Keywords: Attention Deficit/Hyperactivity Disorder; ADHD; Attention Deficit Disorder; ADD; Magnesium
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — threonic acid

ARMS (1):
- L-Threonic Acid Magnesium Salt (L-TAMS) (Experimental): Subjects received open label L-Threonic acid Magnesium salt for 12 weeks. Subjects took MMFS202 (6-hour release) and MMFS302 (12-hour release) by mouth each day, up to three times a day.
  Interventions: Drug: L-Threonic Acid Magnesium Salt (L-TAMS)

INTERVENTIONS:
Drug: L-Threonic Acid Magnesium Salt (L-TAMS)

SUMMARY:
This study is a 12-week, open-label pilot study to test the effects of MMFS-201-301 on cognition and function in adults with ADHD. Subjects may enter the trial on a stable dose of medication for ADHD, and MMFS-201-301 will be given. Subjects who do not enter on a stable dose of ADHD medication will receive MMFS-201-301 alone.

ELIGIBILITY:
Inclusion Criteria:

* Male or female adults ages 18-55 years of age
* A diagnosis of childhood-onset Attention Deficit/Hyperactivity Disorder (ADHD), meeting the Diagnostic and Statistical Manual, Fifth Edition (DSM-V) criteria for ADHD in adulthood, including at least 5 current symptoms of inattentive or impulsive-hyperactive traits, and childhood onset by age 12, defined as two symptoms of inattentive or of impulsive/hyperactive traits by the age of 12
* A score of 20 or more on the Adult ADHD Investigator Symptom Report Scale (AISRS), and, for those individuals stably treated with stimulants, a Clinical Global Impression -ADHD (CGI-ADHD) severity score of no greater than 4 ("moderately ill")
* Subjects on a stable dose of stimulant medication must be treated on the same dose for at least 1 month prior to study entry

Exclusion Criteria:

* A history of intolerance to magnesium supplementation, or the ingredients in MMFS202 (6-hour release) AND MMFS302 (12-hour release)
* Pregnant or nursing females
* A known unstable medical illness including hepatic, renal, gastroenterological, respiratory, cardiovascular (including hypertension ≥ 140/90 mmHg at screening), endocrinologic (e.g. thyroid), neurologic (e.g. seizure), immunologic, hematologic, or psychiatric (other than ADHD) disorder); individuals with kidney dysfunction will be excluded, as dysfunctional kidneys may have difficulty clearing the magnesium from the body (which can result in dangerously high magnesium levels); individuals with heart block will be excluded from the study
* Any medical condition that the Principal Investigator (PI) believes will be exacerbated by study participation
* A history of cancer (except localized skin cancer without metastases or in situ cervical cancer) within 5 years prior to screening
* A known history of narrow-angle glaucoma
* Current (within 3 months) DSM-V criteria for abuse or dependence with any psychoactive substance other than nicotine
* Intelligence Quotient (IQ) less than 80 (based on the Wechsler Abbreviated Scale of Intelligence-II Full Scale IQ calculation)
* Multiple adverse drug reactions
* Any other concomitant medication with primarily central nervous system activity as specified in the study protocol
* Current use of a monoamine-oxidase inhibitor (MAOI) or use within the past two weeks
* Current use of antibiotics, as the study agent may reduce the absorption of antibiotics
* Subjects may not take any of the following substances for at least 7 days prior to baseline and throughout the study: Calcium channel blockers; any psychoactive medications; any medications known to interact with magnesium; supplemental magnesium or any magnesium-containing products; all dietary or herbal supplements or products including those purported to improve memory, improve sleep, or decrease stress.
* Investigator and his/her immediate family; defined as the investigator's spouse, parent, child, grandparent, or grandchild

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2016-03; Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Craig Surman, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- L-Threonic Acid Magnesium Salt (L-TAMS): Subjects took open label L-Threonic acid Magnesium salt for 12 weeks. Subjects took MMFS202 (6-hour release) and MMFS302 (12-hour release) by mouth each day, up to three times a day.
Period: Overall Study
Arm/Group | L-Threonic Acid Magnesium Salt (L-TAMS)
Started | 20 (20 subjects signed consent to participate in the study. 15 subjects began taking L-TAMS.)
Treated | 15
Completed | 13
Not Completed | 7
Not completed — Lost to Follow-up | 2
Not completed — Physician Decision | 1
Not completed — Withdrawal by Subject | 1
Not completed — Screen Fail | 3

BASELINE CHARACTERISTICS:
Population: 15 participants began taking MMFS-201-301 daily.
Arm/Group | L-Threonic Acid Magnesium Salt (L-TAMS)
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 15
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.4 (14.04)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 6
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 4
  White | 9
  More than one race | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 15

OUTCOME MEASURES:

1. Primary Outcome: Change in Adult ADHD Investigator Symptom Rating Scale (AISRS) Score
Description: The Adult ADHD Investigator Symptom Report Scale (AISRS) assesses each of the 18 individual symptoms of ADHD in DSM-IV on a Likert scale from 0 (not present) to 3 (severe), with a total possible score of 54.
  The change in AISRS score from baseline to endpoint (12 weeks) was calculated as the later time point score minus the earlier time point score.
Time Frame: Baseline and 12 Weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | L-Threonic Acid Magnesium Salt (L-TAMS)
Number analyzed (Participants) | 15
units on a scale | -6.3 (8.8)

ADVERSE EVENTS:
Time Frame: Adverse events were collected for the entire time that subjects were exposed to L-TAMS (12 weeks).
Arm/Group | L-Threonic Acid Magnesium Salt (L-TAMS)
All-Cause Mortality (participants affected / at risk) | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 10/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | L-Threonic Acid Magnesium Salt (L-TAMS) (N=15)
Nausea/Vomit/Diarrhea (Gastrointestinal disorders) | 5 (8)
Muscle Discomfort (Musculoskeletal and connective tissue disorders) | 2 (5)
Drooling/Sweating (Nervous system disorders) | 1 (1)
Cold/Infection/Allergy (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Headache (General disorders) | 3 (3)
Dry Skin (Skin and subcutaneous tissue disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Burned Finger (Injury, poisoning and procedural complications) | 1 (1)
Decreased Concentration (Psychiatric disorders) | 1 (1)
Metallic Taste in Mouth (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-05-10): https://cdn.clinicaltrials.gov/large-docs/90/NCT02558790/Prot_SAP_000.pdf